

# BROWN UNIVERSITY CONSENT FOR RESEARCH PARTICIPATION

Effects of Atomoxetine on Adolescent Alcoho Version 6.0, 28SEP2021

We invite you to be part of a research study directed by Dr. Robert Miranda and his associates at Brown University. You were selected as a possible participant in this study because you said you're interested in reducing your alcohol use.

The researchers will explain this study to you. **Research studies are voluntary and include only people who choose to take part.** Please take your time about deciding whether to participate in this study. Before deciding:

- You can discuss this study with your parents.
- You can also discuss it with your health care doctor.
- If you have any questions, you can ask the researchers for more information.

#### **KEY INFORMATION:**

- PURPOSE: This study is about whether the study medicine plus a computerized alcohol education program helps teenagers reduce their alcohol use. **This is not a treatment study.**
- PROCEDURES: You will take a study medication for 6 weeks; answer personal questions, such as questions about drug and alcohol use, both in person and in your daily life using a smartphone; complete medical tests, including an alcohol breathalyzer, physical exam, heart rate, blood pressure, a urine drug and, if female, pregnancy test; provide a blood sample at a local laboratory; go through a task where you look at water and an alcoholic drink and answer questions; and take part in 7 computerized alcohol education sessions.
- TIME INVOLVED: After screening and during the 6-week study, you will attend weekly 30-minute visits; seven 30-minute computerized alcohol education sessions, two 2-hour assessment sessions; one 10-minute phone interview two weeks after you stop the study medication; and two 30-minute phone interviews 3- and 6-months after you finish taking the study medicine.
- COMPENSATION: If you complete the study, you will receive \$510 for your time.
- RISKS: Possible risks include discomfort or bruising with drawing blood; loss of privacy; undue
  influence; discomfort answering personal questions; and side effects of the medication, such as
  nausea, vomiting, fatigue, decreased appetite, abdominal pain, sleepiness or drowsiness,
  constipation, dry mouth, dizziness, erectile dysfunction, and urinary hesitation, severe injury,
  heart-related problems, suicidal thoughts, hearing voices.
- BENEFITS: Alcohol education and the study medication may help you cutback or abstain from alcohol.
- ALTERNATIVES TO PARTICIPATION: We do not offer other options. There are local treatment programs, however, and you will get a list of services.
- REMOTE OPTION: If in-person visits are not possible, we may offer you the option to have some of
  your visits completed remotely, via telephone or Zoom video conference. Parts of the in-person
  visits that cannot be done over the telephone or Zoom video conference may be excluded or
  rescheduled. You may be asked to sign in or download an app to use Brown University's Zoom
  platform for teleconferencing, depending on your device, and you will need WIFI connection.

#### WHY IS THIS STUDY BEING DONE?

This study will test if a medicine called atomoxetine helps young people reduce their alcohol use. Doctors use this drug to treat attention-deficit/hyperactivity disorder (ADHD). We hope it will help youth reduce their drinking. But we don't know this for sure. There is no medicine to help teenagers reduce their alcohol use. This drug appears to reduce alcohol use in adults with ADHD. This study is the first to test its effects on alcohol use among teenagers who want to reduce their drinking.

#### WHAT WILL HAPPEN IF YOU TAKE PART IN THIS STUDY?

# Before you begin the study:

Before you begin this study, we need to find out if this study is right for you. This **screening** <u>takes</u> <u>about 2.5 hours total, sometimes split across two days</u>. You will take an alcohol breath test and if your alcohol level is above 0.00% at any study visit you will need to return another day.

We will ask you questions about your health and alcohol and drug use. You will give urine and blood samples and have a physical exam by a study doctor. We will test urine for illegal drugs and, if female, pregnancy. If your urine is positive for any illegal drug except marijuana, you won't be able to be in the study. Females cannot be in this study if they are pregnant or breastfeeding.

To see if the study is a good fit, what is one thing that you will need to complete?

# **During the study**:

- If you are a good fit for this study, you will come to our office for a **pre-medication session**. You will take an alcohol breath test, urine drug test and, if female, a pregnancy test. You will answer more questions about yourself. We will record your heart rate, blood pressure, and urge to drink alcohol while you relax and while you look at water and an alcoholic drink. This is called a **cue reactivity assessment**. It may take time for your urge to go down. If your urge remains high, you will meet with a study clinician to help manage your craving. This session will take about 2.5 hours.
- You will attend **6 weekly checkup visits** at our office, <u>each lasting about 30 minutes</u>. During these visits, you will complete an alcohol breath test and provide a urine sample to test for drug use and, if female, pregnancy. We will record your blood pressure and heart rate. We will also ask you about side effects, your mood, any new medications or therapy, and recent alcohol and drug use. Once you start the study medicine, you will return any unused capsules and get more.
- You will complete **two telephone interviews** that last about <u>10 minutes each</u>. One happens in Week 1 and one happens two weeks after your last visit in our offices. We'll ask about any side effects, other medication use or counseling, alcohol withdrawal symptoms, and the number of medication capsules you've taken. We'll also remind you about dose increases and your next scheduled visit.
- You will also receive seven brief alcohol education sessions at our offices about your alcohol use, including your thoughts about cutting back, how your drinking compares to others, and how alcohol is harmful. We'll help you track of your drinking and set goals to cut down. One session will occur at the pre-medication session and at each of the 6 weekly checkup visits. These sessions will Everyone will get the alcohol education program regardless of how much they drink. <a href="Each session lasts about 30 minutes">Each session lasts about 30 minutes</a>. If possible, sessions will happen on the same days as your weekly checkups.
- For six weeks, you will take medication capsules that contain atomoxetine or placebo; one capsule per day for the first three days and then two per day thereafter. You'll take the same type of capsule (atomoxetine or placebo) during the wholestudy. About one-half of youth will get the study medicine; the other half will take placebo pills that look like medicine but are not real. Placebo pills should have no physical effect on you. We will use a

method of chance to decide the group you're in (e.g., **medication assignment**). This method is like flipping a coin. You will not know which group you are in. Neither will the researchers. A prescription for the study medicine or placebo will include your name, address, and date of birth.

- Starting in Week 1, you will **use a study smartphone** to answer questions as you go about your daily life for <u>six weeks</u>. You will answer questions when you wake up, drink alcohol, and when it beeps (about 4 times per day). You'll record where you are, what you're doing, how you're feeling, urges to drink, and how many alcoholic drinks you drank (if any). You can shut it off when you're sleeping or can't respond, like when you're driving, operating machinery, or in other situations where it would be unsafe. We'll check in to see how you're doing and answer any questions.
- During the Week 5 checkup, you will do a second cue reactivity assessment just like the first. We'll
  measure your urge to drink alcohol while you relax and while you look at water and an alcoholic
  drink. You will also provide a blood sample at a local laboratory to test the levels of study medicine
  in your blood. This entire visit, combined with the alcohol education session, will take about 2.5
  hours.

# After you finish alcohol education and the study medicine:

You will complete a **final in-clinic visit** after you complete the study medicine(or placebo). This visit takes about 60 minutes. You will also complete two brief **follow-up interviews** over the phone, 3- and 6-months after you finish the study medicine, about your recent alcohol and drug use. Each interview will take <u>about 30 minutes</u>.

Please explain two or three things that will happen if you decide to participate in this study.

#### SCHEDULE OF ASSESSMENTS

| | Screening | Pre-<br>Medication<br>Session | <u>W</u> | eekly<br>2 | | eckuj<br>4 | <u>5 Vi</u><br>5 | sits<br>6 | Final<br>In-Clinic<br>Visit | Two-<br>week<br>Phone<br>Checkup | Follow-up<br>Interviews<br>(3 & 6<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Alcohol breathalyzer | • | • | • | • | • | • | • | • | • | | |
| Blood pressure & heart rate | • | | • | • | • | • | • | • | | | |
| Blood draw | • | | | | | | • | | | | |
| Phone interview (10 min.) | | | • | | | | | | | • | |
| Cue reactivity assessment | | • | | | | | • | | | | |
| Interviews & questionnaires | • | • | • | • | • | • | • | • | • | | |
| Physical Exam | • | | | | | | | | | | |
| Smartphone assessments | | | • | • | • | • | • | • | | | |
| Urine drug test | • | • | • | • | • | • | • | • | • | | |
| Urine pregnancy test | • | • | • | • | • | • | • | • | • | | |
| Phone interview (30 min.) | | | | | | | | | | | • |
| Alcohol education sessions | | • | • | • | • | • | • | • | | | |

#### HOW LONG WOULD YOU BE IN THIS STUDY?

The study takes about 8 weeks plus two brief phone interviews 3- and 6-months after you finish taking the study medicine.

#### WILL YOU BE PAID FOR YOUR PARTICIPATION?

If you complete the study, you will get \$510.00 in gift certificates or using ClinCard (see below). We will pay you for all parts of the study you complete, even if you decide to stop the study early for any reason. The payment schedule will be as follows:

| Screening session | \$20 | |
|---|---|---|
| Blood tests & physical exam | \$20 | |
| Baseline session | \$20 | |
| 6 weekly checkup visits | \$120 | |
| 6-week smartphone period | \$210 | \$5 per day for using the smartphone app |
| Final in-clinic visit | \$20 | |
| Bonus | \$40 | For returning smartphone (if applicable) & remaining capsules |
| 2-week phone checkup | \$20 | |
| 3- and 6-month phone interviews | \$40 | \$20 for each follow-up interview completed |
| | \$510.00 | |

Payment for participating in this study may be made using ClinCard, a pre-paid Mastercard that works like a debit card.

We will give you the card. You will be given one card for the entire time of your participation and this card may be used to pay you in any future Brown University studies that use ClinCard. You will also get information about how to use this card and whom to call if you have any questions. Be sure to read this information, including the cardholder agreement from Greenphire.

Money will be added to your card based on the study's payment schedule. You may use this card online or at any store that accepts Mastercard. Please read the FAQ information sheet from your study coordinator for details about the ways you can use the card, some of which may involve fees that will reduce the amount of money on the card.

If you earn \$600 or more from Brown University in a single calendar year (either in a one study or across multiple studies), Brown will ask for your social security number to correctly identify you in the payment system and send you an IRS 1099 Form. You may also be asked to complete a Form W9. This may affect your taxes. Only payments for being in research studies will be used to decide if you should receive the IRS form. Money for study-related parking, food, and other expenses are not included in this IRS disclosure.

This card is administered by an outside company called Greenphire. Greenphire will be given your name, address, and date of birth. They will use this information only as part of the payment system, and it will not be given or sold to any other company. Greenphire will not receive any information about your health status or the study in which you are participating.

If your card is lost or stolen, please call the study coordinator for a free replacement card. If you request a replacement card from Greenphire directly, you may be charged a fee.

Please note that you do not need to use ClinCard to be in this study. You can chose to receive study payments in gift cards instead.

#### WHAT KINDS OF RISKS OR DISCOMFORTS COULD YOU EXPECT?

#### Known risks and discomforts:

• Study medicine risks: Many studies have researched the effects of atomoxetine in children (ages 6 years and older), teenagers, and adults. Studies show it is safe with teenagers and it does not harmfully interact with alcohol in adults; interactions with alcohol are unknown in adolescents. Adult heavy drinkers, non-heavy drinkers, and non-drinkers tolerate this medicine equally well.

Most Common Side Effects Nausea, vomiting, fatigue, decreased appetite, abdominal pain, somnolence (sleepiness or drowsiness), constipation, dry mouth, dizziness, erectile dysfunction, and urinary hesitation

Less Common Side Effects Insomnia, irritability, decrease in weight, anorexia, headache, increased blood pressure, flushing, mydriasis (pupil dilatation), sinus tachycardia (fast heart beat), asthenia (weakness/loss of strength), palpitations (hard, fast or irregular heartbeats), mood swings, dyspepsia (indigestion), chills, feeling jittery, thirst, paresthesia (tingling, tickling, pricking, numbness or burning feeling on your skin), dysuria (painful urination), dysmenorrhea (painful menstruation), delayed ejaculation/ejaculation disorder, hyperhidrosis (increased sweating/perspiration), hot flush, sedation, chest pain, nervousness

Peripheral coldness, prostatitis (prostate inflammation), testicular pain, abnormal orgasm, flatulence (gas), feeling cold, muscle spasm, dysgeusia (abnormal/change in taste), agitation, restlessness, micturition urgency (frequent or urgent urination), pollakiuria (frequent need to urinate), pruritus (itching), urticarial (hives), flushing, tremor, irregular menstruation, rash, urinary retention, anxiety, diarrhea, back pain, oropharyngeal (mouth) pain, pharyngolaryngeal (pharynx and the larynx) pain, tremor, excoriation (skin scratching), conjunctivitis (pinkeye), syncope (fainting/passing out), blurred vision, panic attacks, hostility, aggressiveness, impulsivity, akathisia (psychomotor restlessness), hypomania, mania

Occasionally, depression and mood problems have been reported and some patients have had suicidal thoughts or actions.

If your mood changes or if you feel depressed or feel you may harm yourself, contact your doctor immediately. Robert Swift, M.D., Ph.D., or Thomas Chun, M.D. (study physicians), Robert Miranda, Ph.D. (clinical psychologist), or another designated licensed mental health professional, will monitor your mood during the study.

Rare But Serious Side Effects Severe liver injury; some signs of liver dysfunction include pruritus (itching), dark urine, jaundice (yellow skin or eyes), right upper stomach tenderness, unexplained flu like symptoms

Heart-related problems, such as sudden death in patients who have heart problems or heart defects, stroke and heart attack in adults, and increased blood pressure and heart rate. Some signs of heart problems include chest pain, shortness of breath, or fainting.

New mental problems in children and teenagers, including suicidal thoughts, psychotic symptoms (e.g., hearing voices, believing things that are not true, being suspicious), or manic symptoms

In males, priapism (painful and nonpainful erection lasting more than 4 hours)

As with any medicine, you may experience an allergic reaction, such as a rash, hives, throat or tongue swelling, shortness of breath, vomiting, lightheadedness or swelling of the lower layer of skin or tissue just under the skin.

#### You should not take atomoxetine if:

- You have an eye problem called narrow angle glaucoma
- You are allergic to anything in atomoxetine (active ingredient: atomoxetine hydrochloride; inactive ingredients: pregelatinized starch, dimethicone, gelatin, sodium laurylsulfate,

FD&C Blue No.2, synthetic yellow iron oxide, titanium dioxide, red iron dioxide, and edible black ink)

o You have or have had a rare tumor called pheochromocytoma.

Before taking atomoxetine **notify us** of all health conditions (or a family history of), especially:

Liver problems High or low blood pressure Depression

Heart problems or defects Psychosis Mental health problems

The study medicine may change how other medications work. So, it is very important to tell us about any new medications you use during the study so we can make sure it's safe. This is especially true if you take medication for asthma, depression, or blood pressure, as well as cold or allergy medicine. You should not take atomoxetine if you have taken an anti-depression medicine called a monoamine oxidase inhibitor or MAOI within the past 14 days. Some names of MAOI medicines are Nardil (phenelzine sulfate), Parnate (tranylcypromine sulfate), and Emsam (selegiline transdermal system).

Be careful driving or using machinery until you know how the medication affects you. It may make you feel sleepy or dizzy, making it hard to drive or perform other activities safely.

- **Placebo risks:** Placebo pills will contain microcrystalline cellulose, a commonly used inactive filler, and 50 mg of riboflavin. Riboflavin is an easily absorbed water-soluble vitamin (B2). There are no known toxic or adverse reactions to riboflavin in humans.
- **Blood draw risks:** Problems drawing blood rarely occur. These include temporary discomfort from the needle stick, local bleeding, a lump or bruising and, rarely, infection, lightheadedness and fainting. Only a small amount of blood will be taken, about 2 teaspoonfuls.
- **Psychological risks:** Some questions we ask may be upsetting or you may feel uncomfortable answering them. If you do not wish to answer a question, you can skip it and go to the next.
- Loss of confidentiality: As this study involves the use of your identifiable, personal information, there is a chance that a loss of confidentiality or privacy will occur. We have procedures in place to reduce the chances of this happening (see "How will information about you and your participation be kept private?" section below).
- **Undue influence:** Undue influence can happen when the payment you get is large. Such pressure is unlikely in this study because payments are fair for the time and effort required and like other studies in the area. There will be no other rewards or payments. Even if you stop, we will pay you for any time you were in the study. If you decide not to participate in this study or decide to stop the study, you will not lose access to needed health services available outside the study.

#### Unknown risks and discomforts:

The study medicine may have side effects that no one knows about yet. The researchers will let you know if they learn of anything that might make you change your mind about participating in this study.

Please explain two or three risks of participating in this study.

# WHO TO CONTACT IF YOU HAVE A STUDY-RELATED INJURY, ILLNESS, OR DISTRESS?

If you get sick or have any problems from taking the study drug you must call your study doctor right away. Dr. Robert Miranda is available during business hours (401-863-6658). Dr. Robert Swift can be reached after hours (401-456-2000); ask to have him paged. We will provide emergency care, if

necessary, but Brown University and the researchers assume no responsibility to pay for such care or to provide financial compensation for emergency or non-emergency health services.

#### ARE THERE ANY BENEFITS IF YOU PARTICIPATE?

You may or may not directly benefit from being in this research study. You will get alcohol education about your alcohol use even if you decide to stop the study medication. You will also have the chance to contribute to research that may be helpful to you or to others in the future.

#### WHAT OTHER CHOICES DO YOU HAVE IF YOU DON'T WANT TO PARTICIPATE?

If you decide not to participate in this study, we do not offer any other study. There are treatment programs in Rhode Island, however, and we will give you a list of those services.

#### HOW WILL INFORMATION ABOUT YOU AND YOUR PARTICIPATION BE KEPT PRIVATE?

# Use of personal information that can identify you:

Any information we collect about you as part of this study that identifies you will remain private. Only a code number will be used to identify your private information; your name will not be matched with your private information. We will keep all information about you locked up and password protected. It will be disclosed only with your permission or as required by law.

Clinical research relies on truthful data collected from you without the fear of disclosure of your sensitive information. Congress authorized the Secretary of Health and Human Services to issue Certificates of Confidentiality that allows research investigators to refuse to disclose identifiable

information about you even under a subpoena. This study has been issued a Certificate of Confidentiality from the National Institute on Alcohol Abuse and Alcoholism (NIAAA). The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you.

The Certificate cannot be used, however, to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects or for information that must be disclosed in order to meet the requirements of the federal FDA.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

As a participant in this study, you must also do your part in protecting your identity and your sensitive information linked to this study: The Certificate of Confidentiality remains protective if you do not disclose your participation to others. Once disclosure is in the public domain, it's possible that the Certificate of Confidentiality can be challenged.

If you give us your permission by signing this document, information, which does not identify you by name, may be used for scientific purposes, including teaching or publication. Because of the investigational nature of this study, the study sponsor, the Brown University Institutional Review Board, the FDA, the Department of Health and Human Services, the Offices of Inspector General and Civil Rights have the right to review study records. Your information will be kept confidential. Your name, address, and date of birth will be used to fill an individualized prescription for atomoxetine or placebo capsules. In addition, for your blood samples to be processed, the laboratory order may include your name, sex at birth and date of birth. We will share this information with the study pharmacy and blood laboratory, when applicable, which adheres to HIPAA practices and stores this information in a private, password-protected, and encrypted format.

# How information about you will be stored:

We maintain all research data and records in a secure location at Brown University. Only authorized individuals will have access to it.

# When will we share some of your private information with others:

Instances when information will not be kept confidential or private involve reports of child abuse, elder abuse, or threats to harm yourself or others. If you report suicidal or homicidal intent or ideation or child or elder abuse, the principal investigator, a clinical psychologist, or study physician will be notified immediately. A report will be filed with the appropriate authorities if abuse is reported.

When are the researchers required to share some of your private information with authorities?

# People and agencies that will have access to your information:

The National Institutes of Health, the Brown University Institutional Review Board, the FDA, the Department of Health and Human Services, the Offices of Inspector General and Civil Rights have the right to review study records.

Members of our research team are part of the Lifespan health system and will have access to the study records. An individual prescription for the study medicine or placebo will include your name, address, and date of birth. We will share this information with the study pharmacy, which adheres to HIPAA practices and stores this information in a private, password-protected, and encrypted format.

#### ARE THERE ANY COSTS FOR TAKING PART IN THIS STUDY?

There will be no cost to you for being in this study.

#### WHAT IF YOU WANT TO STOP PARTICIPATING IN THIS STUDY?

You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time. Refusing to participate in or stop the study will not affect your current or future relationship with Brown University, Dr. Robert Miranda, or other researchers. If you want to stop, it is important to tell us so that we can get any remaining medication and, if applicable, the smartphone device from you.

Can you change your mind and stop your participation in this study?

# WHO CAN YOU CONTACT IF YOU HAVE QUESTIONS ABOUT THIS STUDY?

#### The Research Team:

You may contact Dr. Robert Miranda at 401-863-6658 or by email at Robert\_Miranda\_Jr@brown.edu with any questions or concerns about the research or your participation in this study.

#### Brown University Human Research Protection Program (HRPP):

If you have questions about your rights while taking part in this study, or you have concerns or suggestions about the study and you want to talk to someone other than the researchers, you may contact Brown's HRPP at 401-863-3050 or email them at IRB@Brown.edu.

# WHERE CAN YOU FIND PUBLIC INFORMATION ABOUT THIS STUDY?

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by US Law. This Web site will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in this study. If you have any questions that are not answered in this consent form, ask one of the study staff.

Please answer YES or NO to the following questions: A. Is this document in a language you understand? В. Do you understand the information in this consent form? C. Have you been given enough time to ask questions and talk about the D. Have all your questions been answered to your satisfaction? E. Do you think you received enough information about the study? F. Do you volunteer to be in this study of your own free will and without being pressured by the investigator or study staff? G. Do you know that you can leave the study at any time without giving a reason and with affecting your health care? H. Do you know that your records from this study may be reviewed by the study sponsor and by government authorities? I. Do you know that you cannot be in another study while you are in this study? You must show that you understand what this study involves by correctly answering the five questions included in this form. To sign this consent form, you must also be able to answer "Yes" to questions A-I listed directly above. Please check whether you agree to be re-contacted for future studies and initial. Yes No \_\_\_\_ (Initial) Your signature below shows that you have read and understood the information in this document. The researchers answered your questions to your satisfaction and you agree to volunteer as a research participant for this study. We will give you a copy of this form. Printed Name of Adult Study Participant Signature of Adult Study Participant Date/Time Printed Name of Person Explaining Consent Form Signature of Person Explaining Consent Form Date/Time



# BROWN UNIVERSITY ASSENT FOR RESEARCH PARTICIPATION

#### Effects of Atomoxetine on Adolescent Alcohol Use

Version 6.0, 28SEP2021

We invite you to be part of a research study directed by Dr. Robert Miranda and his associates at Brown University. You were selected as a possible participant in this study because you said you're interested in reducing your alcohol use.

The researchers will explain this study to you. **Research studies are voluntary and include only people who choose to take part.** Please take your time about deciding whether to participate in this study. Before deciding:

- You can discuss this study with your parents.
- You can also discuss it with your health care doctor.
- If you have any questions, you can ask the researchers for more information.

#### **KEY INFORMATION:**

- PURPOSE: This study is about whether the study medicine plus a computerized alcohol education program helps teenagers reduce their alcohol use. **This is not a treatment study.**
- PROCEDURES: You will take a study medication for 6 weeks; answer personal questions, such as questions about drug and alcohol use, both in person and in your daily life using a smartphone; complete medical tests, including an alcohol breathalyzer, physical exam, heart rate, blood pressure, a urine drug and, if female, pregnancy test; provide a blood sample at a local laboratory; go through a task where you look at water and an alcoholic drink and answer questions; and take part in 7 computerized alcohol education sessions. We will also ask your parents some questions about you.
- TIME INVOLVED: After screening and during the 6-week study, you will attend weekly 30-minute visits; seven 30-minute computerized alcohol education sessions, two 2-hour assessment sessions; one 10-minute phone interview two weeks after you stop the study medication; and two 30-minute phone interviews 3- and 6-months after you finish taking the study medicine.
- COMPENSATION: If you complete the study, you will receive \$510 for your time.
- RISKS: Possible risks include discomfort or bruising with drawing blood; loss of privacy; undue
  influence; discomfort answering personal questions; and side effects of the medication, such as
  nausea, vomiting, fatigue, decreased appetite, abdominal pain, sleepiness or drowsiness,
  constipation, dry mouth, dizziness, erectile dysfunction, and urinary hesitation, severe injury,
  heart-related problems, suicidal thoughts, hearing voices.
- BENEFITS: Alcohol education and the study medication may help you cutback or abstain from alcohol.
- ALTERNATIVES TO PARTICIPATION: We do not offer other options. There are local treatment programs, however, and you will get a list of services.
- REMOTE OPTION: If in-person visits are not possible, we may offer you the option to have some of your visits completed remotely, via telephone or Zoom video conference. Parts of the in-person visits that cannot be done over the telephone or Zoom video conference may be excluded or

rescheduled. You may be asked to sign in or download an app to use Brown University's Zoom platform for teleconferencing, depending on your device, and you will need WIFI connection.

#### WHY IS THIS STUDY BEING DONE?

This study will test if a medicine called atomoxetine helps young people reduce their alcohol use. Doctors use this drug to treat attention-deficit/hyperactivity disorder (ADHD). We hope it will help youth reduce their drinking. But we don't know this for sure. There is no medicine to help teenagers reduce their alcohol use. This drug appears to reduce alcohol use in adults with ADHD. This study is the first to test its effects on alcohol use among teenagers who want to reduce their drinking.

#### WHAT WILL HAPPEN IF YOU TAKE PART IN THIS STUDY?

# Before you begin the study:

First, we will ask your parents if they give their permission for you to take part in this study. If they don't agree, you cannot be in this study. If your parents do agree, and you agree too, here is what will happen next.

Before you begin this study, we need to find out if this study is right for you. This **screening** <u>takes</u> <u>about 2.5 hours, sometimes split across two days</u>. You will take an alcohol breath test and if your alcohol level is above 0.00% at any study visit you will need to return another day.

We will ask your parents some questions about you. We will ask you questions about your health and alcohol and drug use. You will give urine and blood samples and have a physical exam by a study doctor. We will test urine for illegal drugs and, if female, pregnancy. If your urine is positive for any illegal drug except marijuana, you won't be able to be in the study. Females cannot be in this study if they are pregnant or breastfeeding. If you decide to participate, your parents will learn about your drinking habits.

To see if the study is a good fit, what is one thing that you will need to complete?

#### During the study:

- If you are a good fit for this study, you will come to our office for a **pre-medication session**. You will take an alcohol breath test, urine drug test and, if female, a pregnancy test. You will answer more questions about yourself. We will record your heart rate, blood pressure, and urge to drink alcohol while you relax and while you look at water and an alcoholic drink. This is called a **cue reactivity assessment**. It may take time for your urge to go down. If your urge remains high, you will meet with a study clinician to help manage your craving. This session will take about 2.5 hours.
- You will attend 6 weekly checkup visits at our office, each lasting about 30 minutes. During these visits, you will complete an alcohol breath test and provide a urine sample to test for drug use and, if female, pregnancy. We will record your blood pressure and heart rate. We will also ask you about side effects, your mood, any new medications or therapy, and recent alcohol and drug use. Once you start the study medicine, you will return any unused capsules and get more.
- You will complete **two telephone interviews** that last about <u>10 minutes each</u>. One happens in Week 1 and one happens two weeks after your last visit in our offices. We'll ask about any side effects, other medication use or counseling, alcohol withdrawal symptoms, and the number of medication capsules you've taken. We'll also remind you about dose increases and your next scheduled visit.
- You will also receive seven brief alcohol education sessions at our offices about your alcohol use, including your thoughts about cutting back, how your drinking compares to others, and how alcohol is harmful. We'll help you track of your drinking and set goals to cut down. One session will occur at the pre-medication session and at each of the 6 weekly checkup visits. Everyone will

get the alcohol education program regardless of how much they drink. <u>Each session lasts about 30</u> minutes. If possible, sessions will happen on the same days as your weekly checkups.

- For six weeks, you will take medication capsules that contain atomoxetine or placebo; one capsule per day for the first three days and then two per day thereafter. You'll take the same type of capsule (atomoxetine or placebo) during the wholestudy. About one-half of youth will get the study medicine; the other half will take placebo pills that look like medicine but are not real. Placebo pills should have no physical effect on you. We will use a method of chance to decide the group you're in (e.g., medication assignment). This method is like flipping a coin. You will not know which group you are in. Neither will the researchers. A prescription for the study medicine or placebo will include your name, address, and date of birth.
- Starting in Week 1, you will **use a study smartphone** to answer questions as you go about your daily life for <u>six weeks</u>. You will answer questions when you wake up, drink alcohol, and when it beeps (about 4 times per day). You'll record where you are, what you're doing, how you're feeling, urges to drink, and how many alcoholic drinks you drank (if any). You can shut it off when you're sleeping or can't respond, like when you're driving, operating machinery, or in other situations where it would be unsafe. We'll check in to see how you're doing and answer any questions.
- During the Week 5 checkup, you will do a second cue reactivity assessment just like the first. We'll
  measure your urge to drink alcohol while you relax and while you look at water and an alcoholic
  drink. You will also provide a blood sample at a local laboratory to test the levels of study medicine
  in your blood. This entire visit, combined with the alcohol education session, will take <u>about 2.5</u>
  hours.

# After you finish alcohol education and the study medicine:

You will complete two brief **follow-up interviews** over the phone, 3- and 6-months after you finish the study medicine, about your recent alcohol and drug use. Each interview will take about 30 minutes.

Please explain two or three things that will happen if you decide to participate in this study.

#### SCHEDULE OF ASSESSMENTS

| | Screening | Pre-<br>Medication<br>Session | | eekly<br>2 | y Cho | eckuj<br>4 | p Vi<br>5 | sits<br>6 | Final<br>In-Clinic<br>Visit | Two-<br>week<br>Phone<br>Checkup | Follow-up<br>Interviews<br>(3 & 6<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Alcohol breathalyzer | • | • | • | • | • | • | • | • | • | | |
| Blood pressure & heart rate | • | | • | • | • | • | • | • | | | |
| Blood draw | • | | | | | | • | | | | |
| Phone interview (10 min.) | | | • | | | | | | | • | |
| Cue reactivity assessment | | • | | | | | • | | | | |
| Interviews & questionnaires | • | • | • | • | • | • | • | • | • | | |
| Physical Exam | • | | | | | | | | | | |
| Smartphone assessments | | | • | • | • | • | • | • | | | |
| Urine drug test | • | • | • | • | • | • | • | • | • | | |
| Urine pregnancy test | • | • | • | • | • | • | • | • | • | | |
| Alcohol education sessions<br>Phone interview (30 min) | | • | • | • | • | • | • | • | | | • |

#### HOW LONG WOULD YOU BE IN THIS STUDY?

The study takes about 8 weeks plus two brief phone interviews 3- and 6-months after you finish taking the study medicine.

#### WILL YOU BE PAID FOR YOUR PARTICIPATION?

If you complete the study, you will get \$510.00 in gift certificates or using ClinCard (see below). We will pay you for all parts of the study you complete, even if you decide to stop the study early for any reason. The payment schedule will be as follows:

| Screening session | \$20 | |
|---|---|---|
| Blood tests & physical exam | \$20 | |
| Baseline session | \$20 | |
| 6 weekly checkup visits | \$120 | |
| 6-week smartphone period | \$210 | \$5 per day for using the smartphone app |
| Final in-clinic visit | \$20 | |
| Bonus | \$40 | For returning smartphone (if applicable) & remaining capsules |
| 2-week phone checkup | \$20 | |
| 3- and 6-month phone interviews | \$40 | \$20 for each follow-up interview completed |
| · | \$510.00 | |

Payment for participating in this study may be made using ClinCard, a pre-paid Mastercard that works like a debit card.

We will give you the card. You will be given one card for the entire time of your participation and this card may be used to pay you in any future Brown University studies that use ClinCard. You will also get information about how to use this card and whom to call if you have any questions. Be sure to read this information, including the cardholder agreement from Greenphire.

Money will be added to your card based on the study's payment schedule. You may use this card online or at any store that accepts Mastercard. Please read the FAQ information sheet from your study coordinator for details about the ways you can use the card, some of which may involve fees that will reduce the amount of money on the card.

If you earn \$600 or more from Brown University in a single calendar year (either in a one study or across multiple studies), Brown will ask for your social security number to correctly identify you in the payment system and send you an IRS 1099 Form. You may also be asked to complete a Form W9. This may affect your taxes. Only payments for being in research studies will be used to decide if you should receive the IRS form. Money for study-related parking, food, and other expenses are not included in this IRS disclosure.

This card is administered by an outside company called Greenphire. Greenphire will be given your name, address, and date of birth. They will use this information only as part of the payment system, and it will not be given or sold to any other company. Greenphire will not receive any information about your health status or the study in which you are participating.

If your card is lost or stolen, please call the study coordinator for a free replacement card. If you request a replacement card from Greenphire directly, you may be charged a fee.

Please note that you do not need to use ClinCard to be in this study. You can chose to receive study payments in gift cards instead.

#### WHAT KINDS OF RISKS OR DISCOMFORTS COULD YOU EXPECT?

#### Known risks and discomforts:

• Study medicine risks: Many studies have researched the effects of atomoxetine in children (ages 6 years and older), teenagers, and adults. Studies show it is safe with teenagers and it does not harmfully interact with alcohol in adults; interactions with alcohol are unknown in adolescents. Adult heavy drinkers, non-heavy drinkers, and non-drinkers tolerate this medicine equally well.

Most Common Side Effects Nausea, vomiting, fatigue, decreased appetite, abdominal pain, somnolence (sleepiness or drowsiness), constipation, dry mouth, dizziness, erectile dysfunction, and urinary hesitation

Less Common Side Effects Insomnia, irritability, decrease in weight, anorexia, headache, increased blood pressure, flushing, mydriasis (pupil dilatation), sinus tachycardia (fast heart beat), asthenia (weakness/loss of strength), palpitations (hard, fast or irregular heartbeats), mood swings, dyspepsia (indigestion), chills, feeling jittery, thirst, paresthesia (tingling, tickling, pricking, numbness or burning feeling on your skin), dysuria (painful urination), dysmenorrhea (painful menstruation), delayed ejaculation/ejaculation disorder, hyperhidrosis (increased sweating/perspiration), hot flush, sedation, chest pain, nervousness.

Peripheral coldness, prostatitis (prostate inflammation), testicular pain, abnormal orgasm, flatulence (gas), feeling cold, muscle spasm, dysgeusia (abnormal/change in taste), agitation, restlessness, micturition urgency (frequent or urgent urination), pollakiuria (frequent need to urinate), pruritus (itching), urticarial (hives), flushing, tremor, irregular menstruation, rash, urinary retention, anxiety, diarrhea, back pain, oropharyngeal (mouth) pain, pharyngolaryngeal (pharynx and the larynx) pain, tremor, excoriation (skin scratching), conjunctivitis (pinkeye), syncope (fainting/passing out), blurred vision, panic attacks, hostility, aggressiveness, impulsivity, akathisia (psychomotor restlessness), hypomania, mania.

Occasionally, depression and mood problems have been reported and some patients have had suicidal thoughts or actions.

If your mood changes or if you feel depressed or feel you may harm yourself, contact your doctor immediately. Robert Swift, M.D., Ph.D., or Thomas Chun, M.D. (study physicians), Robert Miranda, Ph.D. (clinical psychologist), or another designated licensed mental health professional, will monitor your mood during the study.

Rare But Serious Side Effects Severe liver injury; some signs of liver dysfunction include pruritus (itching), dark urine, jaundice (yellow skin or eyes), right upper stomach tenderness, unexplained flu like symptoms.

Heart-related problems, such as sudden death in patients who have heart problems or heart defects, stroke and heart attack in adults, and increased blood pressure and heart rate. Some signs of heart problems include chest pain, shortness of breath, or fainting.

New mental problems in children and teenagers, including suicidal thoughts, psychotic symptoms (e.g., hearing voices, believing things that are not true, being suspicious), or manic symptoms.

In males, priapism (painful and nonpainful erection lasting more than 4 hours).

As with any medicine, you may experience an allergic reaction, such as a rash, hives, throat or tongue swelling, shortness of breath, vomiting, lightheadedness or swelling of the lower layer of skin or tissue just under the skin.

#### You should not take atomoxetine if:

- You have an eye problem called narrow angle glaucoma
- You are allergic to anything in atomoxetine (active ingredient: atomoxetine hydrochloride; inactive ingredients: pregelatinized starch, dimethicone, gelatin, sodium lauryl sulfate, FD&C Blue No.2, synthetic yellow iron oxide, titanium dioxide, red iron dioxide, and edible black ink)
- o You have or have had a rare tumor called pheochromocytoma.

Before taking atomoxetine **notify us** of all health conditions (or a family history of), especially:

Liver problems High or low blood pressure Depression

Heart problems or defects Psychosis Mental health problems

The study medicine may change how other medications work. So, it is very important to tell us about any new medications you use during the study so we can make sure it's safe. This is especially true if you take medication for asthma, depression, or blood pressure, as well as cold or allergy medicine. You should not take atomoxetine if you have taken an anti-depression medicine called a monoamine oxidase inhibitor or MAOI within the past 14 days. Some names of MAOI medicines are Nardil (phenelzine sulfate), Parnate (tranylcypromine sulfate), and Emsam (selegiline transdermal system).

Be careful driving or using machinery until you know how the medication affects you. It may make you feel sleepy or dizzy, making it hard to drive or perform other activities safely.

- **Placebo risks:** Placebo pills will contain microcrystalline cellulose, a commonly used inactive filler, and 50 mg of riboflavin. Riboflavin is an easily absorbed water-soluble vitamin (B2). There are no known toxic or adverse reactions to riboflavin in humans.
- **Blood draw risks:** Problems drawing blood rarely occur. These include temporary discomfort from the needle stick, local bleeding, a lump or bruising and, rarely, infection, lightheadedness and fainting. Only a small amount of blood will be taken, about 2 teaspoonfuls.
- **Psychological risks:** Some questions we ask may be upsetting or you may feel uncomfortable answering them. If you do not wish to answer a question, you can skip it and go to the next.
- Loss of confidentiality: As this study involves the use of your identifiable, personal information, there is a chance that a loss of confidentiality or privacy will occur. We have procedures in place to reduce the chances of this happening (see "How will information about you and your participation be kept private?" section below).
- **Undue influence:** Undue influence can happen when the payment you get is large. Such pressure is unlikely in this study because payments are fair for the time and effort required and like other studies in the area. There will be no other rewards or payments. Even if you stop, we will pay you for any time you were in the study. If you decide not to participate in this study or decide to stop the study, you will not lose access to needed health services available outside the study.

Please explain two or three risks of participating in this study.

#### **Unknown risks and discomforts:**

The study medicine may have side effects that no one knows about yet. The researchers will let you know if they learn of anything that might make you change your mind about participating in this study.

# WHO TO CONTACT IF YOU HAVE A STUDY-RELATED INJURY, ILLNESS, OR DISTRESS?

If you get sick or have any problems from taking the study drug you must call your study doctor right away. Dr. Robert Miranda is available during business hours (401-863-6658). Dr. Robert Swift can be reached after hours (401-456-2000); ask to have him paged. We will provide emergency care, if necessary, but Brown University and the researchers assume no responsibility to pay for such care or to provide financial compensation for emergency or non-emergency health services.

#### ARE THERE ANY BENEFITS IF YOU PARTICIPATE?

You may or may not directly benefit from being in this research study. You will get alcohol education about your alcohol use even if you decide to stop the study medication. You will also have the chance to contribute to research that may be helpful to you or to others in the future.

#### WHAT OTHER CHOICES DO YOU HAVE IF YOU DON'T WANT TO PARTICIPATE?

If you decide not to participate in this study, we do not offer any other study. There are treatment programs in Rhode Island, however, and we will give you a list of those services.

#### HOW WILL INFORMATION ABOUT YOU AND YOUR PARTICIPATION BE KEPT PRIVATE?

#### Use of personal information that can identify you:

Any information we collect about you as part of this study that identifies you will remain private. Only a code number will be used to identify your private information; your name will not be matched with your private information. We will keep all information about you locked up and password protected. It will be disclosed only with you and your parent's permission or as required by law.

To help protect your privacy, we obtained a Certificate of Confidentiality from the National Institutes of Health. With this certificate, we cannot be forced to share information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings.

The Certificate remains protective as long as you do not tell others about your participation.

#### How information about you will be stored:

We maintain all research data and records in a secure location at Brown University. Only authorized individuals will have access to it.

# When will we share some of your private information with others:

If you tell us that someone has hurt you, another child, or an elder person we must tell people who are responsible for protecting children and elders to ensure that everyone is safe. Likewise, if you tell us you are thinking about hurting or killing yourself or someone else, we need to tell people who are responsible for protecting children. This may include your parents.

When are the researchers required to share some of your private information with authorities?

#### People and agencies that will have access to your information:

The National Institutes of Health, the Brown University Institutional Review Board, the FDA, the Department of Health and Human Services, the Offices of Inspector General and Civil Rights have the right to review study records.

Members of our research team are part of the Lifespan health system and will have access to the study records. An individual prescription for the study medicine or placebo will include your name, address, and date of birth. In addition, for your blood samples to be processed, the laboratory order may include your name, sex at birth and date of birth. We will share this information with the study pharmacy and blood laboratory, when applicable, which adheres to HIPAA practices and stores this information in a private, password-protected, and encrypted format.

### ARE THERE ANY COSTS FOR TAKING PART IN THIS STUDY?

There will be no cost to you for being in this study.

#### WHAT IF YOU WANT TO STOP PARTICIPATING IN THIS STUDY?

You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time. In addition, even if your parents say "yes" you can still decide not to do this or change your mind. Refusing to participate in or stop the study will not affect your current or future relationship with Brown University, Dr. Robert Miranda, or other researchers. If you want to stop, it is important to tell us so that we can get any remaining medication and, if applicable, the smartphone device from you.

Can you change your mind and stop your participation in this study?

# WHO CAN YOU CONTACT IF YOU HAVE QUESTIONS ABOUT THIS STUDY?

#### The Research Team:

You may contact Dr. Robert Miranda at 401-863-6658 or by email at Robert\_Miranda\_Jr@brown.edu with any questions or concerns about the research or your participation in this study.

#### Brown University Human Research Protection Program (HRPP):

If you have questions about your rights while taking part in this study, or you have concerns or suggestions about the study and you want to talk to someone other than the researchers, you may contact Brown's HRPP at 401-863-3050 or email them at IRB@Brown.edu.

#### WHERE CAN YOU FIND PUBLIC INFORMATION ABOUT THIS STUDY?

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by US Law. This Web site will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in this study. If you have any questions that are not answered in this consent form, ask one of the study staff.

Please answer YES or NO to the following questions: A. Is this document in a language you understand? В. Do you understand the information in this consent form? C. Have you been given enough time to ask questions and talk about the study? D. Have all your questions been answered to your satisfaction? E. Do you think you received enough information about the study? F. Do you volunteer to be in this study of your own free will and without being pressured by the investigator or study staff? Do you know that you can leave the study at any time without giving a G. reason and with affecting your health care? H. Do you know that your records from this study may be reviewed by the study sponsor and by government authorities? I. Do you know that you cannot be in another study while you are in this study? You must show that you understand what this study involves by correctly answering the five questions included in this form. To sign this consent form, you must also be able to answer "Yes" to questions A-I listed directly above. Please check whether you agree to be re-contacted for future studies and initial. Yes No (Initial) Your signature below shows that you have read and understood the information in this document. The researchers answered your questions to your satisfaction and you agree to volunteer as a research participant for this study. We will give you a copy of this form. Printed Name of Minor (< 18 years old) Study Participant Signature of Minor (< 18 years old) Study Participant Date/Time Printed Name of Person Explaining Assent Form Signature of Person Explaining Assent Form Date/Time



# BROWN UNIVERSITY PARENT PERMISSION FOR RESEARCH PARTICIPATION OF MINOR

# Effects of Atomoxetine on Adolescent Alcohol Use

Version 6.0, 28SEP2021

Dr. Robert Miranda and his associates at Brown University are conducting a research study. Your child was selected as a possible participant in this study because they expressed interest in reducing their alcohol use. Your child's **participation in this research study is voluntary**.

The researchers will explain this study to you. Please take your time to decide whether to allow your child to participate in this study. Before deciding:

- You can discuss this study with your child.
- You can also discuss it with your child's health care doctor.
- If you have any questions, you can ask the researchers for more information.

#### **KEY INFORMATION:**

- PURPOSE: This study is about whether the study medicine plus a computerized alcohol education program helps teenagers reduce their alcohol use. **This is not a treatment study.**
- PROCEDURES: Your child will take a study medication for 6 weeks; answer personal questions, such as questions about drug and alcohol use, both in person and in their daily life using a smartphone; complete medical tests, including an alcohol breathalyzer, physical exam, heart rate, blood pressure, a urine drug and, if female, pregnancy test; provide a blood sample at a local laboratory; complete a task where they look at water and an alcoholic drink and answer questions; and take part in 7 computerized alcohol education sessions. We will also ask you some questions about your child.
- TIME INVOLVED: After screening and during the 6-week study, your child will attend weekly 30-minute visits; seven 30-minute computerized alcohol education; two 2-hour assessment sessions; one 10-minute phone interview two weeks after they stop the study medication; and two 30-minute phone interviews 3- and 6-months after they finish taking the study medicine.
- COMPENSATION: If your child completes the study, they will receive \$510 for their time.
- RISKS: Possible risks include discomfort or bruising with drawing blood; loss of privacy; undue
  influence; discomfort answering personal questions; and side effects of the medication, such as
  nausea, vomiting, fatigue, decreased appetite, abdominal pain, sleepiness or drowsiness,
  constipation, dry mouth, dizziness, erectile dysfunction, and urinary hesitation, severe injury,
  heart-related problems, suicidal thoughts, hearing voices.
- BENEFITS: Alcohol education and the study medication may help your child cutback or abstain from alcohol.
- ALTERNATIVES TO PARTICIPATION: We do not offer other options. There are local treatment programs, however, and you and your child will get a list of services.
- REMOTE OPTION: If in-person visits are not possible, we may offer your child the option to have some of their visits completed remotely, via telephone or Zoom video conference. Parts of the inperson visits that cannot be done over the telephone or Zoom video conference may be excluded or rescheduled. They may be asked to sign in or download an app to use Brown University's Zoom platform for teleconferencing, depending on your device, and they will need WIFI connection.

#### WHY IS THIS STUDY BEING DONE?

This study will test if a medicine called atomoxetine helps young people reduce their alcohol use. Doctors use this drug to treat attention-deficit/hyperactivity disorder (ADHD). We hope it will help youth reduce their drinking. But we don't know this for sure. There is no medicine to help teenagers reduce their alcohol use. This drug appears to reduce alcohol use in adults with ADHD. This study is the first to test its effects on alcohol use among teenagers who want to reduce their drinking.

#### WHAT WILL HAPPEN IF YOUR CHILD TAKES PART IN THIS STUDY?

# Before your child begins the study:

First, we will ask your permission for your child to take part in this study. If you don't agree, your child cannot be in this study. If you do agree, and your child agrees too, here is what will happen next.

Before your child begins this study, we need to find out if this study is right for them. This **screening** takes about 2.5 hours, sometimes split across two days. Your child will take an alcohol breath test and if their alcohol level is above 0.00% at any study visit they will need to return another day.

We will ask you some questions about your child. We will ask your child questions about their health and alcohol and drug use. Your child will give urine and blood samples and have a physical exam by a study doctor. We will test urine for illegal drugs and, if female, pregnancy. If their urine is positive for any illegal drug except marijuana, your child won't be able to be in the study. Females cannot be in this study if they are pregnant or breastfeeding.

To see if the study is a good fit, what is one thing that your child will need to complete?

# **During the study**:

- If your child is a good fit for this study, they will come to our office for a **pre-medication session**. They will take an alcohol breath test, urine drug test and, if female, a pregnancy test. Your child will answer more questions about himself or herself. We will record their heart rate, blood pressure, and urge to drink alcohol while they relax and while they look at water and an alcoholic drink. This is called a **cue reactivity assessment**. It may take time for their urge to go down. If their urge remains high, they will meet with a study clinician to help manage their craving. This session will take about 2.5 hours.
- He or she will attend **6 weekly checkup visits** at our office, <u>each lasting about 30 minutes</u>. During these visits, they will complete an alcohol breath test and provide a urine sample to test for drug use and, if female, pregnancy. We will record their blood pressure and heart rate. We will also ask them about side effects, their mood, any new medications or therapy, and recent alcohol and drug use. Once they start the study medicine, they will return any unused capsules and get more.
- He or she will complete two telephone interviews that last about 10 minutes each. One happens in
  Week 1 and one happens two weeks after their last visit in our offices. We'll ask about any side
  effects, other medication use or counseling, alcohol withdrawal symptoms, and the number of
  medication capsules they've taken. We'll also remind them about dose increases and their next
  scheduled visit.
- He or she will also receive **seven brief alcohol education sessions** about their alcohol use, including their thoughts about cutting back, how their drinking compares to others, and how alcohol is harmful. We'll help them track of their drinking and set goals to cut down. One session will occur at the pre-medication session and at each of the 6 weekly checkup visits. Everyone will get the alcohol education program regardless of how much they drink. <u>Each session lasts about 30 minutes</u>. If possible, sessions will happen on the same days as their weekly checkups.

- For six weeks, he or she will take medication capsules that contain atomoxetine or placebo; one capsule per day for the first three days and then two per day thereafter. They'll take the same type of capsule (atomoxetine or placebo) during the wholestudy. About one-half of youth will get the study medicine; the other half will take placebo pills that look like medicine but are not real. Placebo pills should have no physical effect on them. We will use a method of chance to decide the group they're in (e.g., medication assignment). This method is like flipping a coin. They will not know which group they're are in. Neither will the researchers. A prescription for the study medicine or placebo will include their name, address, and date of birth.
- Starting in Week 1, they will **use a study smartphone** to answer questions as they go about their daily life for <u>six weeks</u>. They'll answer questions when they wake up, drink alcohol, and when it beeps (about 4 times per day). They'll record where they are, what they're doing, how they're feeling, urges to drink, and how many alcoholic drinks they drank (if any). They can shut it off when they're sleeping or can't respond, like when they're driving, operating machinery, or in other situations where it would be unsafe. We'll check in to see how they're doing and answer any questions.
- During the Week 5 checkup, they will do a second **cue reactivity assessment** just like the first. We'll measure their urge to drink alcohol while they relax and look at water and an alcoholic drink. They will also provide a blood sample at a local laboratory to test the levels of study medicine in their blood. This entire visit, combined with the alcohol education session, will take about 2.5 hours.

# After you finish alcohol education and the study medicine:

He or she will complete two brief **follow-up interviews** over the phone, 3 and 6 months after they finish the study medicine, about their recent alcohol and drug use. Each will take <u>about 30 minutes</u>.

Please explain two or three things that will happen if your child participates in this study.

#### SCHEDULE OF ASSESSMENTS

| | Screening | Pre-<br>Medication<br>Session | | eekly<br>2 | | eckuj<br>4 | <u>o Vi</u><br>5 | sits<br>6 | Final<br>In-Clinic<br>Visit | Two-<br>week<br>Phone<br>Checkup | Follow-up<br>Interviews<br>(3 & 6<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Alcohol breathalyzer | • | • | • | • | • | • | • | • | • | | |
| Blood pressure & heart rate | • | | • | • | • | • | • | • | | | |
| Blood draw | • | | | | | | • | | | | |
| Phone interview (10 min.) | | | • | | | | | | | • | |
| Cue reactivity assessment | | • | | | | | • | | | | |
| Interviews & questionnaires | • | • | • | • | • | • | • | • | • | | |
| Physical Exam | • | | | | | | | | | | |
| Smartphone assessments | | | • | • | • | • | • | • | | | |
| Urine drug test | • | • | • | • | • | • | • | • | • | | |
| Urine pregnancy test | • | • | • | • | • | • | • | • | • | | |
| Phone interview (30 min.) | | | | | | | | | | | • |
| Alcohol education sessions | | • | • | • | • | • | • | • | | | |

#### HOW LONG WOULD YOUR CHILD BE IN THIS STUDY?

The study takes about 8 weeks plus two brief phone interviews 3- and 6-months after he or she finishes taking the study medicine.

#### WILL YOUR CHILD BE PAID FOR HIS OR HER PARTICIPATION?

If your child completes the study, they will get \$510.00 in gift certificates or using ClinCard (see below). We will pay them for all parts of the study they complete, even if they decide to stop the study early for any reason. The payment schedule will be as follows:

| Screening session | \$20 | |
|---|---|---|
| Blood tests & physical exam | \$20 | |
| Baseline session | \$20 | |
| 6 weekly checkup visits | \$120 | |
| 6-week smartphone period | \$210 | \$5 per day for using the smartphone app |
| Final in-clinic visit | \$20 | |
| Bonus | \$40 | For returning smartphone (if applicable) & remaining capsules |
| 2-week phone checkup | \$20 | |
| 3- and 6-month phone interviews | \$40 | \$20 for each follow-up interview completed |
| | \$510.00 | |

Payment for participating in this study may be made using ClinCard, a pre-paid Mastercard that works like a debit card.

We will give your child the card. They will be given one card for the entire time of their participation and this card may be used to pay them in any future Brown University studies that use ClinCard. They will also get information about how to use this card and whom to call if they have any questions. Be sure to read this information, including the cardholder agreement from Greenphire.

Money will be added to their card based on the study's payment schedule. They may use this card online or at any store that accepts Mastercard. Please read the FAQ information sheet from the study coordinator for details about the ways they can use the card, some of which may involve fees that will reduce the amount of money on the card.

If your child earns \$600 or more from Brown University in a single calendar year (either in a one study or across multiple studies), Brown will ask for their social security number to correctly identify them in the payment system and send them an IRS 1099 Form. They may also be asked to complete a Form W9. This may affect their taxes. Only payments for being in research studies will be used to decide if they should receive the IRS form. Money for study-related parking, food, and other expenses are not included in this IRS disclosure.

This card is administered by an outside company called Greenphire. Greenphire will be given your child's name, address, and date of birth. They will use this information only as part of the payment system, and it will not be given or sold to any other company. Greenphire will not receive any information about your child's health status or the study in which they are participating.

If their card is lost or stolen, please call the study coordinator for a free replacement card. If they request a replacement card from Greenphire directly, they may be charged a fee.

Please note that your child does not need to use ClinCard to be in this study. They can chose to receive study payments in gift cards instead.

# WHAT KINDS OF RISKS OR DISCOMFORTS COULD YOU EXPECT?

#### Known risks and discomforts:

• **Study medicine risks:** Many studies have researched the effects of atomoxetine in children (ages 6 years and older), teenagers, and adults. Studies show it is safe with teenagers and it does not

harmfully interact with alcohol in adults; interactions with alcohol are unknown in adolescents. Adult heavy drinkers, non-heavy drinkers, and non-drinkers tolerate this medicine equally well.

Most Common Side Effects Nausea, vomiting, fatigue, decreased appetite, abdominal pain, somnolence (sleepiness or drowsiness), constipation, dry mouth, dizziness, erectile dysfunction, and urinary hesitation

Less Common Side Effects Insomnia, irritability, decrease in weight, anorexia, headache, increased blood pressure, flushing, mydriasis (pupil dilatation), sinus tachycardia (fast heart beat), asthenia (weakness/loss of strength), palpitations (hard, fast or irregular heartbeats), mood swings, dyspepsia (indigestion), chills, feeling jittery, thirst, paresthesia (tingling, tickling, pricking, numbness or burning feeling on your skin), dysuria (painful urination), dysmenorrhea (painful menstruation), delayed ejaculation/ejaculation disorder, hyperhidrosis (increased sweating/perspiration), hot flush, sedation, chest pain, nervousness.

Peripheral coldness, prostatitis (prostate inflammation), testicular pain, abnormal orgasm, flatulence (gas), feeling cold, muscle spasm, dysgeusia (abnormal/change in taste), agitation, restlessness, micturition urgency (frequent or urgent urination), pollakiuria (frequent need to urinate), pruritus (itching), urticarial (hives), flushing, tremor, irregular menstruation, rash, urinary retention, anxiety, diarrhea, back pain, oropharyngeal (mouth) pain, pharyngolaryngeal (pharynx and the larynx) pain, tremor, excoriation (skin scratching), conjunctivitis (pinkeye), syncope (fainting/passing out), blurred vision, panic attacks, hostility, aggressiveness, impulsivity, akathisia (psychomotor restlessness), hypomania, mania.

Occasionally, depression and mood problems have been reported and some patients have had suicidal thoughts or actions.

If your mood changes or if you feel depressed or feel you may harm yourself, contact your doctor immediately. Robert Swift, M.D., Ph.D., or Thomas Chun, M.D. (study physicians), Robert Miranda, Ph.D. (clinical psychologist), or another designated licensed mental health professional, will monitor your mood during the study.

Rare But Serious Side Effects Severe liver injury; some signs of liver dysfunction include pruritus (itching), dark urine, jaundice (yellow skin or eyes), right upper stomach tenderness, unexplained flu like symptoms.

Heart-related problems, such as sudden death in patients who have heart problems or heart defects, stroke and heart attack in adults, and increased blood pressure and heart rate. Some signs of heart problems include chest pain, shortness of breath, or fainting.

New mental problems in children and teenagers, including suicidal thoughts, psychotic symptoms (e.g., hearing voices, believing things that are not true, being suspicious), or manic symptoms.

In males, priapism (painful and nonpainful erection lasting more than 4 hours).

As with any medicine, your child may experience an allergic reaction, such as a rash, hives, throat or tongue swelling, shortness of breath, vomiting, lightheadedness or swelling of the lower layer of skin or tissue just under the skin.

# Your child should not take atomoxetine if:

o He or she has an eye problem called narrow angle glaucoma

- He or she is allergic to anything in atomoxetine (active ingredient: atomoxetine hydrochloride; inactive ingredients: pregelatinized starch, dimethicone, gelatin, sodium lauryl sulfate, FD&C Blue No.2, synthetic yellow iron oxide, titanium dioxide, red iron dioxide, and edible black ink)
- o He or she has or has had a rare tumor called pheochromocytoma.

Before taking atomoxetine **notify us** of all health conditions (or a family history of), especially:

Liver problems High or low blood pressure Depression

Heart problems or defects Psychosis Mental health problems

The study medicine may change how other medications work. So, it is very important to tell us about any new medications your child uses during the study so we can make sure it's safe. This is especially true if your child takes medication for asthma, depression, or blood pressure, as well as cold or allergy medicine. Your child should not take atomoxetine if they have taken an anti-depression medicine called a monoamine oxidase inhibitor or MAOI within the past 14 days. Some names of MAOI medicines are Nardil (phenelzine sulfate), Parnate (tranylcypromine sulfate), and Emsam (selegiline transdermal system).

Your child should be careful driving or using machinery until they know how the medication affects them. It may make them feel sleepy or dizzy, making it hard to drive or perform other activities safely.

- **Placebo risks:** Placebo pills will contain microcrystalline cellulose, a commonly used inactive filler, and 50 mg of riboflavin. Riboflavin is an easily absorbed water-soluble vitamin (B2). There are no known toxic or adverse reactions to riboflavin in humans.
- **Blood draw risks:** Problems drawing blood rarely occur. These include temporary discomfort from the needle stick, local bleeding, a lump or bruising and, rarely, infection, lightheadedness and fainting. Only a small amount of blood will be taken, about 2 teaspoonfuls.
- **Psychological risks:** Some questions we ask may be upsetting or your child may feel uncomfortable answering them. If they do not wish to answer a question, they can skip it and go to thenext.
- Loss of confidentiality: As this study involves the use of your child's identifiable, personal information, there is a chance that a loss of confidentiality or privacy will occur. We have procedures in place to reduce the chances of this happening (see "How will information about you and your participation be kept private?" section below).
- **Undue influence:** Undue influence can happen when the payment a child gets is large. Such pressure is unlikely in this study because payments are fair for the time and effort required and like other studies in the area. There will be no other rewards or payments. Even if your child stops, we will pay them for any time they were in the study. If your child decides not to participate in this study or decides to stop the study, they will not lose access to needed health services available outside the study.

Please explain two or three risks of participating in this study.

#### Unknown risks and discomforts:

The study medicine may have side effects that no one knows about yet. The researchers will let you and your child know if they learn of anything that might make you or your child change your mind about participating in this study.

#### WHO TO CONTACT IF YOU HAVE A STUDY-RELATED INJURY, ILLNESS, OR DISTRESS?

If your child gets sick or has any problems from taking the study drug you or your child must call your study doctor right away. Dr. Robert Miranda is available during business hours (401-863-6658). Dr. Robert Swift can be reached after hours (401-456-2000); ask to have him paged. We will provide emergency care, if necessary, but Brown University and the researchers assume no responsibility to pay for such care or to provide financial compensation for emergency or non-emergency health services.

#### ARE THERE ANY BENEFITS IF YOU PARTICIPATE?

Your child may or may not directly benefit from being in this research study. Your child will get alcohol education about their alcohol use even if they decide to stop the study medication. They will also have the chance to contribute to research that may be helpful to them or to others in the future.

# WHAT OTHER CHOICES DO YOU HAVE IF YOU DON'T WANT TO PARTICIPATE?

If you decide not to allow your child to participate in this study, we do not offer any other study. There are treatment programs in Rhode Island, however, and we will give you and your child a list of those services.

# HOW WILL INFORMATION ABOUT YOU AND YOUR PARTICIPATION BE KEPT PRIVATE?

# Use of personal information that can identify you:

Any information we collect about your child as part of this study that identifies them will remain private. Only a code number will be used to identify your child's private information; their name will not be matched with their private information. We will keep all information about them locked up and password protected. It will be disclosed only with you and your child's permission or as required by law.

Clinical research relies on truthful data collected from your child without the fear of disclosure of their sensitive information. Congress authorized the Secretary of Health and Human Services to issue Certificates of Confidentiality that allows research investigators to refuse to disclose identifiable information about your child even under a subpoena. This study has been issued a Certificate of Confidentiality from the National Institute on Alcohol Abuse and Alcoholism (NIAAA). The researchers can use this Certificate to legally refuse to disclose information that may identify your child in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify them.

The Certificate cannot be used, however, to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects or for information that must be disclosed in order to meet the requirements of the federal FDA.

You and your child should understand that a Certificate of Confidentiality does not prevent you or your child from voluntarily releasing information about himself or herself or their involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

As a participant in this study, your child must also do their part in protecting their identity and their sensitive information linked to this study: The Certificate of Confidentiality remains protective if they do not disclose their participation to others. Once disclosure is in the public domain, it's possible that the Certificate of Confidentiality can be challenged.

If you give us your permission by signing this document, information, which does not identify your child by name, may be used for scientific purposes, including teaching or publication. Because of the investigational nature of this study, the study sponsor, the Brown University Institutional Review Board, the FDA, the Department of Health and Human Services, the Offices of Inspector General and

Civil Rights have the right to review study records. Your child's information will be kept confidential. His or her name, address, and date of birth will be used to fill an individualized prescription for atomoxetine or placebo capsules. In addition, for your child's blood samples to be processed, the laboratory order may include their name, sex at birth and date of birth. We will share this information with the study pharmacy and blood laboratory, when applicable, which adheres to HIPAA practices and stores this information in a private, password-protected, and encrypted format.

# How information about you will be stored:

We maintain all research data and records in a secure location at Brown University. Only authorized individuals will have access to it.

# When will we share some of your private information with others:

If your child tells us that someone has hurt them, another child, or an elder person we must tell people who are responsible for protecting children and elders to ensure that everyone is safe. Likewise, if your child tells us he or she are thinking about hurting or killing himself/herself or someone else, we need to tell people who are responsible for protecting children. This may include telling you.

When are the researchers required to share some of your child's private information with authorities?

# People and agencies that will have access to your information:

The National Institutes of Health, the Brown University Institutional Review Board, the FDA, the Department of Health and Human Services, the Offices of Inspector General and Civil Rights have the right to review study records.

Members of our research team are part of the Lifespan health system and will have access to the study records. An individual prescription for the study medicine or placebo will include your child's name, address, and date of birth. We will share this information with the study pharmacy, which adheres to HIPAA practices and stores this information in a private, password-protected, and encrypted format.

#### ARE THERE ANY COSTS FOR TAKING PART IN THIS STUDY?

There will be no cost to you or your child for being in this study.

# WHAT IF YOU WANT TO STOP PARTICIPATING IN THIS STUDY?

Your child does not have to be in this study if you or they do not want them to be. Even if you give permission for them to be in this study, you can change your mind and stop at any time. In addition, even if you say "yes" your child can still decide not to do this or change his or her mind. Refusing to participate in or stop the study will not affect you or your child's current or future relationship with Brown University, Dr. Robert Miranda, or other researchers. If your child wants to stop, it is important to tell us so that we can get any remaining medication and, if applicable, the smartphone device from them.

Can your child change his or her mind and stop participating in this study?

#### WHO CAN YOU CONTACT IF YOU HAVE QUESTIONS ABOUT THIS STUDY?

# The Research Team:

You or your child may contact Dr. Robert Miranda at 401-863-6658 or by email at Robert\_Miranda\_Jr@brown.edu with any questions or concerns about the research or your child's participation in this study.

# Brown University Human Research Protection Program (HRPP):

If you have questions about your rights while your child is taking part in this study, or you have concerns or suggestions about the study and you want to talk to someone other than the researchers, you may contact Brown's HRPP at 401-863-3050 or email them at IRB@Brown.edu.

# WHERE CAN YOU FIND PUBLIC INFORMATION ABOUT THIS STUDY?

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by US Law. This Web site will not include information that can identify your child. At most, the website will include a summary of the results. You can search this website at any time.

# AGREEMENT FOR YOUR CHILD TO BE IN THE STUDY

This parent permission form contains important information to help you decide if you want your child to be in this study. If you have any questions that are not answered in this parent permission form, ask one of the study staff.

Please answer YES or NO to the following questions:

| A. | Is this document in a language you understand? | |
|---|---|---|
| В. | Do you understand the information in this parent permission form? | |
| C. | Have you been given enough time to ask questions and talk about the study? | he |
| D. | Have all your questions been answered to your satisfaction? | <del>.</del> |
| E. | Do you think you received enough information about the study? | |
| F. | Do you give permission for your child to be in this study of your ow<br>will and without being pressured by the investigator or study staff? | |
| G. | Do you know that your child can leave the study at any time without a reason and with affecting his or her health care? | ut giving |
| H. | Do you know that your child's records from this study may be reviet<br>the study sponsor and by government authorities? | ewed by |
| I. | Do you know that your child cannot be in another study while you this study? | are in |
| | se check whether you agree we can re-contact your child for future s Yes No (Initial) | tudies and initial. |
| | t Name of Child | |
| Prin | ted Name of Parent/Legal Guardian | |
| Sigr | ature of Parent/Legal Guardian | Date/Time |
| Prin<br>Fori | ted Name of Person Explaining Parent/Legal Guardian Permission<br>n | |
| Sigr<br>Fori | ature of Person Explaining Parent/Legal Guardian Permission | Date/Time |